CLINICAL TRIAL: NCT07365553
Title: Omega-3 Fatty Acids and Autism Spectrum Disorder (ASD) - A Double-blind Randomized Controlled Trial of Omega-3 Fatty Acids in Youth With ASD
Brief Title: Omega-3, Autism Spectrum Disorder (ASD)
Acronym: OMeASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Pei-Chen Chang, PI, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH110-REC3-113
Record Dates: First submitted 2024-05-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: ASD
Keywords: inflammation; adolescent; omega-3
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: To investigate the effects of DHA, EPA and placebo in adolescents with ASD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega-3 (EPA) (Experimental): EPA
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): Soybean Oil
  Interventions: Dietary Supplement: Placebo
- Omega-3 (DHA) (Experimental): DHA
  Interventions: Dietary Supplement: Omega-3

INTERVENTIONS:
Dietary Supplement: Omega-3 — Omega-3 PUFAs
  Arms: Omega-3 (DHA); Omega-3 (EPA)
Dietary Supplement: Placebo — Soybean Oil
  Arms: Placebo

SUMMARY:
This is a 12 week study to investigate the effects of omega-3 polyunsaturated fatty acids (PUFAs) in youth with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
This is a 12 week study to investigate the effects of omega-3 PUFAs in children (6-17 years-old) with ASD.

The primary outcome will be the clinical symptoms rated by the Aberrant Behavior Checklist (ABC). The secondary outcomes will be inflammatory biomarkers, cognitive function and physiological markers such as heart-rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DSM5 ASD made by child and adolescent psychiatrist
* age 6-17 years-old at the time of enrolment
* no pharmacotherapy or non-pharmacotherapy adjustment within the past 4 weeks,
* Signed informed consent.

Exclusion Criteria:

* comorbid other psychiatric disorders, including schizophrenia or affective mood disorder (Bipolar and Major Depressive Disorder), or substance use disorder
* comorbid physical disorders, such as thyroid dysfunction, cerebral palsy, coagulation disorders
* currently using omega-3 supplements or probiotics
* allergy to omega-3.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Symptoms-Behavioral problems (Aberrant Behavior Checklist, ABC) | Baseline, week 1,2,4,8,12
  The ABC will be used to assess the behavioral problems of participants. It consists of 58 items that describe various behaviors, such as aggression or hyperactivity, and is typically completed by a caregiver or teacher who knows the individual well. Each item is rated on a 4-point scale: 0 = not at all a problem, 1 = slight problem, 2 = moderate problem, and 3 = severe problem. Scores are summed across all items to produce a total score ranging from 0 to 174, with higher scores indicating more severe or frequent problem behaviors

SECONDARY OUTCOMES:
Concentration of blood inflammatory biomarkers in pg/mL | Baseline and week 12
  Interleukin (IL)-1 beta (picogram/milliliter, pg/ML) IL-6 IL-10 Tumor necrosis factor -αlpha Interferon (IFN)-γ
Cognitive function-attention and impulsivity (Continuous Performance Test, CPT) | Baseline and week 12
  CPT will be used to measure the attention and impulsivity in the subjects.
Clinical symptoms: Behavioral problems (Strength and Difficulty Questionnaire, SDQ) | Baseline and week 12
  SDQ will be used to assess behavior problems of the participants. SDQ is a brief behavioral screening tool for children and adolescents, typically aged 3-16, designed to assess emotional and behavioral difficulties as well as prosocial strengths. It has 25 items divided into five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Problems, and Prosocial Behavior, with each subscale containing 5 items. Items are rated on a 3-point scale: 0 = "Not True," 1 = "Somewhat True," 2 = "Certainly True." Scoring involves summing the first four subscales to calculate a Total Difficulties Score (range 0-40), while the Prosocial subscale is scored separately (range 0-10) as a measure of strengths. Higher Total Difficulties Scores indicate greater behavioral or emotional problems, while higher Prosocial scores indicate stronger social skills.
Stool Sample | Baseline and week 12
  Gut microbiomal sequencing, Faecal short-chain fatty acids
Heart Rate variability (HRV) | Baseline and week 12
  Autonomic nervous function (ANS) will be assessed with HRV.
Concentration of blood high-sensitivity C-reactive Protein (hs-CRP) | Baseline and week 12
  measurement of peripheral blood hs-CRP units in milligram/Liter (mg/L)
Concentration of Red Blood Cell (RBC) Polyunsaturated Fatty Acids (PUFAs) | Baseline and week 12
  Measurement of RBC PUFAs units in %
Cognitive function: memory (Wechsler Memory Scale, WMS) | Baseline and week 12
  WMS will be used to measure memory function of the subjects.
Clinical symptoms: attention and hyperactivity (Swanson, Nolan, and Pelham Rating Scale - Version IV, SNAP-IV) | Baseline and week 12
  The SNAP-IV is used to assess attention, hyperactivity and oppositional defiant disorder symptoms in the subjects. It contains 26 items rated on a 4-point scale from 0 ("Not at all") to 3 ("Very much"), reflecting the frequency or severity of each behavior. The items are grouped into three subscales: Inattention, Hyperactivity/Impulsivity, and Oppositional Defiant behaviors, with scores summed within each subscale. Higher scores indicate more severe symptoms, and the scale can be completed by parents, teachers, or clinicians to provide a reliable measure for both clinical evaluation and research.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chen Chang, MD, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No